CLINICAL TRIAL: NCT06826469
Title: The Efficacy and Safety of Task-state-based Temporal Interference Stimulation (TI) in the Treatment of Patients With Depression
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20240117C-R1
Record Dates: First submitted 2024-09-29; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Temporal Interference Stimulation (Experimental): Specific electrode sites are customized for the subject through magnetic resonance scanning, the deep nucleus cluster to be stimulated-nucleus accumbens is calibrated through electric field simulation before treatment, and the stimulation target can be accurately positioned by stimulating the specific electrode sites of the subject during treatment.
  Interventions: Device: Temporal Interference Stimulation

INTERVENTIONS:
Device: Temporal Interference Stimulation — During the treatment period, all subjects were treated with a fixed time interference stimulation (TI) device at a frequency of 30 minutes twice a day, 5 days a week, for a total of 10 treatments. The output current intensity during treatment is 3.64 mA+4.36 mA.

SUMMARY:
This study intends to investigate the intervention efficacy of temporal interference stimulation (TI) on mood symptoms in depressed patients, as well as to explore the neuroimaging mechanisms of TI improvement in depressed patients using pre- and post-treatment magnetic resonance.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-50 years old, right-handed, and completed nine years of compulsory education;
2. Met Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnostic criteria for depression;
3. HAMD-17≥18;
4. Subject was a first-time medication-naïve patient or had previously used antidepressant medication and was currently off medication for ≥2 weeks;
5. The subject/ legal guardian is willing to actively cooperate with the treatment and sign an informed consent form after fully understanding the temporal interference stimulus (TI).

Exclusion Criteria:

1. Co-morbid other psychiatric disorders, including bipolar disorder, affective psychiatric disorders, anxiety spectrum disorders, mental retardation, substance dependence (abuse), etc.;
2. Severe suicidal ideation or behavior;
3. History of a serious physical illness or a disease that may affect the central nervous system;
4. Neurologic disorders or risk of seizures such as previous cranial disorders, head trauma, abnormal electroencephalograms, magnetic resonance evidence of structural brain abnormalities, or a family history of epilepsy;
5. Contraindications to magnetic resonance scanning or time-interference stimulation (TI), such as the presence of metallic or electronic devices in the body (intracranial metallic foreign bodies, cochlear implants, pacemakers and stents, and other metallic foreign bodies);
6. Those who have received or are receiving electroconvulsive therapy (ECT ), modified electroconvulsive therapy (MECT ), transcranial magnetic stimulation (TMS), transcranial direct current stimulation (tDCS), transcranial alternating current stimulation (tACS), or other neurostimulation treatments;
7. Pregnant and lactating women, and women of childbearing age with positive urine pregnancy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Scale（HAMD-17) | 0-5 days
  The Hamilton Depression Scale（HAMD-17) was used to assess the extent of the patient's depressive episodes, with higher scores representing more severe depression, and this scale was used to monitor the patient's improvement in depression before and after treatment.

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale（MADRS） | 0-5 days
  The Montgomery-Asberg Depression Rating Scale (MADRS) is used to reflect the effectiveness of antidepressant treatment and to monitor changes in a patient's condition. The scale is a stand-alone scale whose ratings are based on a clinical interview with questioning about symptoms that leads to a rating of depression severity.
Beck Scale for Suicide Ideation (BSS) | 0-5 days
  The Beck Suicidal Ideation Scale was used to assess the patients' suicidal ideation.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No